CLINICAL TRIAL: NCT01117870
Title: Randomized, Placebo Controlled, Double-blinded Trial to Assess the Effectiveness of Pulse RadioFrequency Treatment of Dorsal Root Ganglion in Patients With Chronic Lumbar Radicular Pain
Brief Title: Assess the Effectiveness of Pulse RadioFrequency in Patients With Chronic Lumbar Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Canadian Pain Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRF-1
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Chronic Pain; Back Pain
Keywords: chronic; pain; lumbar; Radicular
MeSH Terms: conditions — Chronic Pain; Back Pain; Bronchiolitis Obliterans Syndrome; Pain | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The needle will be continuously stimulated at a low voltage to give a sensation of PRF treatment.
  Interventions: Other: Placebo
- Pulsed Radiofrequency (Experimental): PRF will be applied for 120 seconds at 42 degrees celsius.
  Interventions: Other: Pulsed Radiofrequency

INTERVENTIONS:
Other: Pulsed Radiofrequency — 120 seconds at 42 degrees celsius
  Arms: Pulsed Radiofrequency
Other: Placebo — Needle will be continuously stimulated at a low voltage to give a sensation of PRF application.
  Arms: Placebo

SUMMARY:
Pulsed RadioFrequency (PRF) is a relatively new technique derived from a well established and proven intervention, thermal radiofrequency (RF). Both procedures are used in the treatment of chronic pain. Unlike RF treatment, PRF does no direct damage to the nerve. During PRF treatment, electrical energy is applied with a small needle to the affected nerve using a pulsed time cycle that delivers short bursts of RF current. This study is interested in looking at the efficacy of PRF for chronic lumbar radicular pain (CLR) and to assess whether a larger scale clinical study with the same methods can be used.

DETAILED DESCRIPTION:
Methodology and Techniques:

Patients would be screened at St Joseph-East End Pain Clinic for Chronic Lumbar Radiculopathy (CLR) of at least 4 months duration. Based on the history and clinical examination, a diagnosis of CLR involving one or more spinal segments is made and noted. The patient is considered eligible for the study if a CT or MRI of lumbar spine done within the last 4 months demonstrates pathology that is concordant with the patient's clinical symptoms. The spinal level(s) targeted for treatment will be based on clinical findings, e.g. if a patient exhibits signs and symptoms of right L4 radiculopathy, and the MRI demonstrates right paracentral disc herniations at both L4-5 and L5-S1, only the L4 DRG will be targeted.

Patients fulfilling the inclusion criteria will be fully explained about the nature of study, interventions involved and the possible complications after which an informed consent will be taken. Enrolled patients would be randomized-according to the method chosen and included in the study according to previously randomized order. He/she will also meet the ASSESSOR (blind to intervention)-who would note down the baseline parameters of the patient and also collect a baseline Oswestry Score chart, along with noting down other parameters.

A patient having bilateral radiculopathy will be treated for his most affected side in the trial. A patient having CLR of more than one segment on one side shall be treated for all the involved segments with the same technique and counted as a single procedure or intervention for the study.

All OR (operating room) personnel, including the physician performing intervention and patient shall be blind to the randomization and treatment. The grouping code, hence the actual treatment will only be known by the person operating the RF machine.

Only the RF technician shall be in view of the working details of the RF machine and the noise of the machine is cut off. This ensures blinding of all involved except the RF technician. After checking for informed consent and other safety checklist, patient will only be revealed as belonging to group A or B.

All interventions will be done as day care procedures in the OR. Patients would continue to use their medications as before. If the pain relief obtained necessitates decrease in the usage of medications that shall be recorded. Similarly unsatisfactory pain relief obtained necessitating increase in the dose or change of medications shall be recorded. The other parameters to be used for statistical analysis are collected as mentioned in the data analysis paragraph.

The patient will have an established IV access. He would be put in prone position. The involved area of back would be made sterile using chlorohexidine 2% and draped. The patient would be connected to continuous monitoring of 3 lead ECG, NIBP (Non-Invasive Blood Pressure) and pulse oximetry. Sedation, if used will be minimal (Grade I or II) to obtain the necessary response of the patient. Under fluoroscopy guidance- particular spinal segment(s) affected is (are) identified and confirmed. LA using 2% lidocaine is infiltrated to the skin at entry site. For both groups a RF needle (Bayliss: 22-G needle, 5-mm curved active tip and 10 cm) is used. With an appropriate fluoroscopy view needle is inserted to the target location in both the groups.

Target location: the DRG which is an enlargement formed by the dorsal nerve root just proximal to its junction with the spinal nerve lies within the dural sleeve and occupies the upper, medial part of the intervertebral foramen (22). It is confirmed with an anteroposterior fluoroscopy view in which it is advanced, if required, until the tip is located one-third to halfway into the pedicle column (18).

Target Confirmation (Malik et al): Appropriate fluoroscopic placement of needle-near DRG at the lumbar area is noted; on anteroposterior x-ray projection, the DRG is described to lie immediately behind the lateral aspect of the facet column at all spinal levels and on lateral x-ray projection, it is localized to the dorsocranial quadrant of the IVF (intervertebral foramen) Proximity of the needle to the DRG is determined by appropriate sensory stimulation with 50 Hz, at more than 0.4 V (avoids intraganglionic placement) and less than or equal to 0.6 V; motor stimulation at 2 Hz with threshold 1.5-2 times greater than sensory threshold to avoid placement near the anterior nerve root. A radiculogram done also confirms the appropriate placement and helps recognise intradural placement of the needle.

Both the groups will have their respective DRG stimulated for sensory confirmation.

Treatment: Once positioned the physician shall indicate to the RF technician as "treatment" only, at which time either PRF or placebo (only continuing sensory stimulation at a low frequency is applied), without revealing.

Application of Intervention: In Group A-PRF; PRF would be applied for 120 seconds at 42 degree centigrade. Group B-placebo; the needle would be continuously stimulated at a low voltage to give a sensation of PRF application and also to obtain the necessary noise to blind the patients.

Only lidocaine 1% 0.5 ml shall be given in both groups before carrying out the treatment.

In both groups the same procedure is done at all the involved spinal segmental levels. After the procedure the patient is shifted to recovery area to be monitored, observed and managed for any side effects. The observer, blind to the interventions, will record the pain scores and also check for side effects observed before the patient is discharged home.

Blinding and Bias control In our study we plan to blind the patient, the treating physician and the assessor for the actual intervention being done. The randomization code, hence the actual treatment will only be known and administered by the person operating the RF machine. The randomization will be concealed in sealed envelopes

Blinding of patients will be achieved by:

Randomization: Patients will be randomly allocated to each group using a 1:1 ratio. The allocation will be blocked using block sizes of 2, 4, 6.

Both interventions will be similarly, including the use of fluoroscopy. Both interventions will be done using the same kind of needle and technique of stimulation.

Patients belonging to placebo group will have a continuous low voltage stimulation to mask the effect of "no intervention".

Blinding of assessor will be achieved by:

Will not know the randomization order, Will not be present during the intervention, Will not be able to access any written or dictated notes regarding the intervention.

Blinding of the treating Physician will be achieved by:

Will not know the randomization order or grouping of patients, Will not be revealed the treatment applied.

Duration of treatment period Treatment intervention period will involve approximately 30 mins to 60 mins of actual intervention done in the OR.

Duration and Frequency of follow up The duration of follow up will be 3 months after the intervention. The frequency of follow up will be as follows,

The patient would be assessed post-intervention on the following days:

1. 30 minutes post-procedure in recovery
2. 24 hrs after-by a phone call (only VAS and side effects)
3. At 1 week post-procedure-Visit to Observer (VAS, ODI, medications, side effects)
4. At 4 weeks post-procedure-Visit to Observer -assessment for success (VAS, ODI, medications, side effects).
5. At 2 months post-procedure-Visit to Observer (VAS, ODI, medications, side effects)
6. At 3 months post -procedure-Visit to Observer-last follow up visit (VAS, ODI, medications, side effects)

Sample Size, Recruitment Rate:

Sample size has been determined based on feasibility considerations. Total duration of recruitment planned is 8 months The proposed target is recruitment for 8 months, with an expectation of 4 patients/month, making a total of 32 patients for the study.

Potential to recruit patients, as 4 patients every month has been calculated based on the TransForaminal Steroid Injections (TFESI) performed in the last 3-6 months and also booked for the next 3-6 months (calculated as monthly) at St Joseph's Healthcare; data obtained from St Joseph's Healthcare Department of Anesthesia and Pain Dept Secretary Office.

TFESI represents a well accepted, presently performed intervention for patients of CLR and most patients suitable for that are potential recruits for this study.

Statistical Tests The Characteristics of the trial participants will be described using mean (standard deviation) or counts as appropriate. We will use a flow diagram to summarize the flow of patients in the trial.

Feasibility outcomes will be reported as counts (proportions).

Duration of The Trial The proposed study would only recruit patients for 8 months and compare with the expected estimation of the recruitment.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* CLR for at least 4 months of more, with concordant findings on either MRI and CT scan
* VAS score of at least 60/100 at presentation
* informed consent

Exclusion Criteria:

* < 18 years of age
* patient refusal
* any contraindication to neuraxial injection such as coagulation disturbance, anticoagulant therapy, bleeding disorder, or infection at site of injection
* anatomical deformity or derangement, either congenital or surgical such as: extreme scoliosis, previous implant or instrumentation making it difficult to access the foramen as evidence by MRI, CT, or plain x-rays
* uncontrolled diabetes or severe coronary vascular disease necessitating continuation of anticoagulation therapy
* known history of psychiatric illness-such as depression or psychosis
* presence of cancer accounting for present symptoms
* patient's inability of communicate in English and inability to understand and fill out the required follow-up questionnaire and form
* allergy to local anesthetics or steroid or contrast medium
* any patient with a history of acute neurological weakness or neurodeficit in the affected limb in terms of measurable motor weakness or abnormal reflexes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Shanthanna, MD, Principal Investigator — St. Joseph's Healthcare Hamilton; Philip Chan, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- East End Clinic, St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shanthanna H, Chan P, McChesney J, Paul J, Thabane L. Assessing the effectiveness of 'pulse radiofrequency treatment of dorsal root ganglion' in patients with chronic lumbar radicular pain: study protocol for a randomized control trial. Trials. 2012 Apr 28;13:52. doi: 10.1186/1745-6215-13-52. PMID 22540851

RESULTS

PARTICIPANT FLOW:
Groups:
- PRF Treatment: PRF will be applied for 120 seconds at 42 degrees celsius.
  Pulsed RadioFrequency: 120 seconds at 42 degrees celsius
Period: Overall Study
Arm/Group | Placebo | PRF Treatment
Started | 15 | 16
Completed | 14 (One did not receive the allocated intervention; (degenerate spine/inability to place needle).) | 16
Not Completed | 1 | 0
Not completed — Inability to place needle | 1 | 0

BASELINE CHARACTERISTICS:
Population: Adult population both male and female >=18 years old
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PRF Treatment | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Full Range); unit: years] | 57.8 [34 to 83] | 63.8 [48 to 85] | 59.5 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Expected recruitment is at least 4 patients per month. At least 80% of eligible patients fulfilling the selection criteria can be recruited. The final assessment was at the end of 15 months, at which time all the subjects were enrolled. Participants withdrawing within 4 weeks after the interventional shall not be included in the study. However participants withdrawing after 4 weeks of the intervention shall be included in the final analysis, on intention to treat principle.
Time Frame: 15 month point
Population: Patients with suspected leg pain were initially approached by the research assistant. Further screening for eligibility was done in the presence of the physician. Suitable patients met with the research assistant (blind to intervention), who noted down the baseline parameters of the patient after obtaining an informed consent.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: Patients meeting eligibility criteria
Arm/Group | Eligible Patients
Number analyzed (Participants) | 41
Participants | 32

2. Primary Outcome: Number of Participants Lost to Follow-up at 3 Months
Description: Patients who were lost to follow-up at 3 months were recorded.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Lost to Follow-up Patients: Patients who were lost to follow-up at 3 months
Arm/Group | Lost to Follow-up Patients
Number analyzed (Participants) | 32
Participants | 3

3. Secondary Outcome: Change in Mean Visual Analogue Scale (VAS) Scores From Baseline to 4 Weeks
Description: Secondary outcomes were considered as exploratory. Is PRF an effective treatment for patients with CLR pain? It will be measured by a change in VAS scores from baseline measurement at recruitment.
  Visual analog scale (VAS) - For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10) on a 10-cm scale.
Time Frame: baseline (at recruitment) and at 4 Weeks
Population: Intent to treat analysis was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: The needle will be continuously stimulated at a low voltage to give a sensation of PRF treatment.
  Placebo: Needle will be continuously stimulated at a low voltage to give a sensation of PRF application.
  The study of the efficacy of cervical PRF-DRG showed significant results favoring PRF-DRG for a 20% pain reduction in VAS score. It has been noted that a 30% reduction in pain appears to reflect at least a moderate clinically important difference, and this needs to be considered in clinical trials.
- PRF Treatment: PRF will be applied for 120 seconds at 42 degrees celsius.
  Pulsed RadioFrequency: 120 seconds at 42 degrees celsius
  The study of the efficacy of cervical PRF-DRG showed significant results favoring PRF-DRG for a 20% pain reduction in VAS score. It has been noted that a 30% reduction in pain appears to reflect at least a moderate clinically important difference, and this needs to be considered in clinical trials.
Arm/Group | Placebo | PRF Treatment
Number analyzed (Participants) | 15 | 16
units on a scale | -5.43 (1.95) | -5.07 (3.01)

4. Secondary Outcome: Assessment of Side Effects
Description: Percentage of patients having side effects after PRF treatment assessed at 1 week compared to placebo group. Assessment of persisting side effects, percentage of patients having side effects after PRF treatment beyond 1 week compared to the placebo group. Side effects could be nausea, headache, momentary increase in pain, fever, tingling, itching, and/or burning skin at point of treatment
Time Frame: 1 week and up to 3 months
Population: Assessment of persisting side effects and percentage of patients having side effects after PRF treatment beyond 1 week compared to the placebo group. Side effects could be nausea, headache, momentary increase in pain, fever, tingling, itching, and/or burning skin at point of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PRF Treatment
Number analyzed (Participants) | 15 | 16
percentage of participants
  % of participants with short term side effects | 0 | 0
  % of participants with persisting side effects | 0 | 0

5. Secondary Outcome: Change in Oswestry Disability Index (ODI) From Baseline to 4 Week
Description: ODI is an index derived from the Oswestry Low Back Pain Questionnaire used to quantify disability for low back pain. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to: care for oneself, walk, sit, sexual function, stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Time Frame: baseline (at recruitment) and at 4 weeks
Population: Success defined as at least 50% improvement in Oswestry Disability Index (ODI) - measured at 4 weeks compared to placebo group.
Measure: Mean (Standard Deviation); unit: percentage change of ODI
Arm/Group | Placebo | PRF Treatment
Number analyzed (Participants) | 15 | 16
percentage change of ODI | -46 (14) | -44 (17)

6. Secondary Outcome: Number of Participants Who Discontinued Analgesics After Intervention
Description: Number of PRF treatment patients with increase or decrease in medication use (either in dose, frequency, or no use), compared with the placebo group.
Time Frame: 4 weeks
Population: Number of participants who discontinued analgesics after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PRF Treatment
Number analyzed (Participants) | 15 | 16
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 4 weeks, 3 months
Arm/Group | Placebo | PRF Treatment
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes